CLINICAL TRIAL: NCT03755271
Title: Hemodynamic Monitoring in Obstetrics
Status: Completed | Type: Observational
Sponsor: University of Catania (Other)
Collaborators: Marinella Astuto (Unknown); Carmelo Minardi (Unknown); Mirko Mineri (Unknown); Francesco Vasile (Unknown); Gaetano Joseph Palumbo (Unknown)
Responsible Party: Principal Investigator, Paolo Murabito, Assistant Professor, University of Catania
Other Study IDs: 1/2018/PO
Record Dates: First submitted 2018-11-19; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Hypotension
Keywords: Intraoperative hypotension; Caesarean section; Spinal anesthesia
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spinal anesthesia has long been considered the first choice technique in caesarean section, but although it is a reliable and safe procedure, it is in some cases associated with undesirable effects. Maternal hypotension after sub-arachnoid anesthesia is a reduction in systolic blood pressure below 100 mmHg or a decrease of 20% compared to baseline values. According to some authors, maternal hypotension occurs up to 80% in women undergoing caesarean section after spinal anesthesia. In order to reduce the incidence of maternal hypotension, some measures can be taken:

* a reduction of aorto-caval compression by manual displacement of the uterus on the left;
* hemodynamic monitoring;
* administration of fluids;
* optimization of the dosage of the local anesthetic;
* use of vasopressors.

The main objective of the study is to investigate, through the use of a continuous non-invasive hemodynamic monitoring system (Clearsight® - Edwards Lifesciences), the incidence of hypotension in pregnant women at risk undergoing spinal anesthesia due to elective cesarean section.

DETAILED DESCRIPTION:
In this prospective observational not-for profit study, 128 patients will be enrolled to measure the incidence of hypotension during spinal anesthesia for elective cesarean section. On the occasion of the preoperative visit, all patients to be subjected to elective cesarean section will be subjected to the Postural Change Test (PCT), a predictive test for maternal hypotension during spinal anesthesia that evaluate changes in heart rate of pregnant women following postural changes. Specifically, after monitoring the heart rate in the supine position, the patient is asked to change decubitus (from supine to left lateral and then back to supine). The test is positive if the patient's heart rate changes more than 10% from baseline.

Once arrived in the obstetric emergency department, parturients with positive Postural Change Test will be subjected to cannulation of a peripheral vein through a 18-20 Gauge needle cannula and the Clearsight hemodynamic monitoring system will be placed on a finger. The investigators will then proceed to the detection of the following parameters:

* Mean Blood Pressure (MAP);
* Heart Rate (HR);
* Stroke volume (SV);
* Stroke volume Index (SVI);
* Cardiac Index (CI). These data will be collected and reported in the data sheet of the study, at different time points (T0 - T9). Basal values will be collected at T0 and T1: at T0 when the patient is in the supine position and at T1 when the patient is in a lateral position. The investigators will then proceed to the administration of a crystalloid bolus (10 ml/kg) and to the execution of spinal anesthesia (T2). The spinal block needle will be inserted, compatibly to the patient's anatomical conditions, at the L3-L4 / L4-L5 spaces. 0.5% hyperbaric Bupivacaine (5 mg/ml) will be administered at a dose depending on the patient's weight and height.

Once the spinal block has been performed, the patient will be immediately placed in a supine position. The investigators will then continue monitoring the parameters listed above using Clearsight® (SV, SVI, MAP, CI) at 2-minute intervals in the phases following spinal anesthesia:

* T3: 2 minutes after spinal anesthesia,
* T4: 4 minutes after spinal anesthesia,
* T5: 6 minutes after spinal anesthesia,
* T6: 8 minutes after spinal anesthesia. The other measurements will be made at skin incision (T7), uterine incision (T8) and extraction (T9).

Any hemodynamic changes (MAP <60 mmHg or CI <2.5), under volemic optimization conditions, will be treated by administration of vasoconstrictors (Etilefrine, intravenous bolus of 1-3 mg).

At the afterbirth, the investigators will proceed to the infusion of liquids and uterotonic according regimens in use at the unit of Anesthesia and Intensive Care of the Universitary Hospital "G. Rodolico" of Catania.

Given the descriptive nature of the study, a formal calculation of the sample size was not made. As secondary end-points, the Stroke Volume variation following spinal anesthesia, the amount of fluids administered, the vasoconstrictor doses used, diuresis, the Apgar index and the fetal pH will be measured. The number of hypotension episodes not detected by the traditional blood pressure monitoring system but detected by the Clearsight system will also be recorded. For the qualitative variables, the absolute frequencies and the percentage frequencies will be calculated. For the quantitative variables, if with normal distribution, mean and standard deviation will be calculated; if with not normal distribution, median and interquartile range will be calculated.

The normality of the distribution will be evaluated through the Kolmogorov-Smirnoff test.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* American Society of Anesthesiologists (ASA) Classification I-II
* Positive Postural Change Test (PCT)
* Signature of informed consent

Exclusion Criteria:

* Age less than 18 years or above 40 years
* American Society of Anesthesiologists (ASA) Classification III-V
* Negative Postural Change Test (PCT)
* Refusal by the parturients to sign the informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 148 pregnant women, at risk of developing hypotension, undergoing spinal anesthesia for elective Caesarean section at the Universitary Hospital "G. Rodolico" of Catania
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension assessed through the use of the non-invasive hemodynamic monitoring system ClearSight | Intraoperatively

SECONDARY OUTCOMES:
Modifications of Stroke Volume (SV) from basal | 2 minutes after spinal anesthesia
Modifications of Stroke Volume (SV) from basal | 4 minutes after spinal anesthesia
Modifications of Stroke Volume (SV) from basal | 6 minutes after spinal anesthesia
Modifications of Stroke Volume (SV) from basal | 8 minutes after spinal anesthesia
Modifications of Stroke Volume (SV) from basal | 2 minutes after cutaneous incision
Modifications of Stroke Volume (SV) from basal | 2 minutes after uterine incision
Modifications of Stroke Volume (SV) from basal | 2 minutes after extraction
Modifications of Stroke Volume Index (SVI) from basal | 2 minutes after spinal anesthesia
Modifications of Stroke Volume Index (SVI) from basal | 4 minutes after spinal anesthesia
Modifications of Stroke Volume Index (SVI) from basal | 6 minutes after spinal anesthesia
Modifications of Stroke Volume Index (SVI) from basal | 8 minutes after spinal anesthesia
Modifications of Stroke Volume Index (SVI) from basal | 2 minutes after cutaneous incision
Modifications of Stroke Volume Index (SVI) from basal | 2 minutes after uterine incision
Modifications of Stroke Volume Index (SVI) from basal | 2 minutes after extraction
Modifications of Cardiac Index (CI) from basal | 2 minutes after spinal anesthesia
Modifications of Cardiac Index (CI) from basal | 4 minutes after spinal anesthesia
Modifications of Cardiac Index (CI) from basal | 6 minutes after spinal anesthesia
Modifications of Cardiac Index (CI) from basal | 8 minutes after spinal anesthesia
Modifications of Cardiac Index (CI) from basal | 2 minutes after cutaneous incision
Modifications of Cardiac Index (CI) from basal | 2 minutes after uterine incision
Modifications of Cardiac Index (CI) from basal | 2 minutes after extraction
Need for inotropes and / or vasopressor during surgery | Intraoperatively
  Doses of inotropes and / or vasopressor administered during surgery
Need for fluids administration during surgery | Intraoperatively
  Volume of fluids administered during surgery for the eventual treatment of hypotension
Volume of urine excreted during surgery | Intraoperatively
Evaluation of fetal health through Apgar score | At 1 and at 5 minute after birth
  The Apgar score is determined by evaluating the newborn baby on five simple criteria (skin color, pulse rate, reflex irritability grimace, activity and respiratory effort) on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. The test is done at 1 and 5 minutes after birth and may be repeated later if the score is and remains low. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts.
Number of hypotension episodes not detected by the traditional pressure cuff but detected by the Clearsight system | Intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Murabito, MD, Principal Investigator — University of Catania; Marinella Astuto, MD, Study Director — University of Catania
Locations (1):
- "G. Rodolico" Presidium of the Azienda Ospedaliero Universitaria "Policlinico-Vittorio Emanuele", Catania, Italy